CLINICAL TRIAL: NCT00915499
Title: Is Adaptive Servo-Ventilation Therapeutically More Effective Than Continuous Positive Airway Pressure In Treating Complex Sleep Apnea Syndrome?
Brief Title: Complex Sleep Apnea Syndrome (CompSAS) Resolution Study
Acronym: CompSAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA-01-08
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Results first posted 2013-02-22 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Complex Sleep Apnea Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASV mode (Active Comparator)
  Interventions: Device: VPAP Adapt SV
- CPAP mode (Active Comparator)
  Interventions: Device: VPAP Adapt SV

INTERVENTIONS:
Device: VPAP Adapt SV — Comparison of ASV and CPAP modes

SUMMARY:
The purpose of this study is to determine whether adaptive servo-ventilation (ASV) or continuous positive airway pressure (CPAP) is better at treating complex sleep apnea over time.

DETAILED DESCRIPTION:
Between 3 and 19% of patients with clinical and polysomnographic features of obstructive sleep apnea syndrome (OSA) develop a high-frequency of central apneas and/or disruptive Cheyne-Stokes respiratory syndrome after application of continuous positive airway pressure (CPAP), a pattern called the complex sleep apnea syndrome (CompSAS). The trial seeks to determine the efficacy of the ASV vs. CPAP modes for the treatment of CompSAS over time. Baseline clinical and laboratory data will be collected, patients will be randomized to one of the two treatments. Overall study participation is approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of complex sleep apnea syndrome (CompSAS)
* Naive to PAP therapy
* Requires CPAP ≤15 cm H2O

Exclusion Criteria:

* Requires supplemental oxygen or with a baseline SaO2 <90%
* Requires CPAP > 15 cm H2O
* Primary diagnosis of moderate to severe chronic obstructive pulmonary disease, neuromuscular disease, chronic hyperventilation, stroke, cognitive impairment, such that could impair ability to answer subjective questions (study questionnaires) or unstable heart failure
* Any contraindication for nasal or oro-nasal positive airway pressure, such as claustrophobia, severe nasal obstruction, or impaired mental status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-05; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy I Morgenthaler, MD, Principal Investigator — Mayo Sleep Disorders Center
Locations (6):
- United States (6):
  - REM Medical, Phoenix, Arizona
  - Northwestern University, Chicago, Illinois
  - NorthShore University Health System, Skokie, Illinois
  - Mayo Center for Sleep Medicine, Mayo Clinic, Rochester, Minnesota
  - Center for Sleep Medicine, Lafayette Hill, Pennsylvania
  - SleepMed of South Carolina, Columbia, South Carolina

REFERENCES:
- [Derived] Morgenthaler TI, Kuzniar TJ, Wolfe LF, Willes L, McLain WC 3rd, Goldberg R. The complex sleep apnea resolution study: a prospective randomized controlled trial of continuous positive airway pressure versus adaptive servoventilation therapy. Sleep. 2014 May 1;37(5):927-34. doi: 10.5665/sleep.3662. PMID 24790271

RESULTS

PARTICIPANT FLOW:
Groups:
- ASV Mode; CPAP Mode: VPAP Adapt SV : Comparison of ASV and CPAP modes for the treatment of complex sleep apnea
Period: Overall Study
Arm/Group | ASV Mode | CPAP Mode
Started | 33 | 33
Completed | 29 | 31
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ASV Mode | CPAP Mode | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 22 | 46
  >=65 years | 9 | 11 | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 59.1 (14.2) | 59.4 (11.7) | 59.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 26 | 30 | 56
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Apnea-hypopnea Index (AHI) Per Polysomnography (PSG) at the End of Treatment Period
Description: AHI refers to the number of apneas and hypopneas that occurred per hour of sleep
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: AHI (events/hour)
Groups:
- ASV Mode: Positive airway pressure in the adaptive servo-ventilation (ASV) mode
- CPAP Mode: Positive airway pressure in the continuous positive airway pressure (CPAP) mode
Arm/Group | ASV Mode | CPAP Mode
Number analyzed (Participants) | 29 | 31
AHI (events/hour) | 4.4 (9.6) | 9.9 (11.1)

2. Secondary Outcome: Quality of Life Measured by the Sleep Apnea Quality of Life Index (SAQLI)
Description: Likert scale measured from 0-7. The minimum important difference a change of 0.5 when a 7-item Likert scale is used. 0 represents the most negative response, 7 represents the most positive response.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ASV Mode | CPAP Mode
Number analyzed (Participants) | 30 | 31
units on a scale
  Baseline SAQLI score | 4.6 (1.2) | 4.5 (0.9)
  End of study SAQLI score | 4.7 (0.9) | 4.6 (1.1)

ADVERSE EVENTS:
Arm/Group | ASV Mode | CPAP Mode
Serious Adverse Events (participants affected / at risk) | 0/33 | 3/33
Other Adverse Events (participants affected / at risk) | 8/33 | 9/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASV Mode (N=33) | CPAP Mode (N=33)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Heart attack (Cardiac disorders) | 0 (0) | 1 (1)
Rebound hypertension (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASV Mode (N=33) | CPAP Mode (N=33)
Facial irritation/rash (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Skin breakdown (from mask) (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Other sinus issues (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less